CLINICAL TRIAL: NCT04401280
Title: Effectiveness of Novel Bioactive Glass in the Treatment of Enamel White Spot Lesions : A Randomized Controlled Trial
Brief Title: Bioactive Glass in the Treatment of Enamel White Spot Lesions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rania Salah (Other)
Collaborators: Queen Mary University of London (Other)
Responsible Party: Sponsor-Investigator, Rania Salah, Clinical instructor and Principal investigator at conservative dentistry department, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WSL treatment
Record Dates: First submitted 2020-05-15; First posted 2020-05-26 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: White Spot Lesion of Tooth
Keywords: Bioactive glass; CPP-ACP; Remineralization; White spot lesions
MeSH Terms: interventions — NovaMin; casein phosphopeptide-amorphous calcium phosphate nanocomplex

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- BiominF® (Active Comparator): Test group
  Interventions: Drug: BiominF
- Novamin® (Active Comparator): Test group
  Interventions: Drug: Novamin
- CPP-ACP (Active Comparator): Control group
  Interventions: Drug: CPP-ACP

INTERVENTIONS:
Drug: BiominF — in office application of bioactive glass followed by self administered application by the patient until a point of white spot remineralization is reached
  Arms: BiominF®
Drug: Novamin — in office application of bioactive glass followed by self administered application by the patient until a point of white spot remineralization is reached
  Arms: Novamin®
Drug: CPP-ACP — applied in accordance with the manufacturer's specifications
  Arms: CPP-ACP

SUMMARY:
the aim of this study is to evaluate the effectiveness of BiominF® and Novamin® in comparison to Casein phosphopeptide-amorphous calcium phosphate (CPP-ACP) in the treatment of enamel white spot lesions

ELIGIBILITY:
Inclusion Criteria:

* Not less than 1 white spot lesion on the labial surface of teeth in the anterior region with code 2 International Caries Detection and Assessment System II (ICDAS-II) or less
* Absence of any active periodontal disease.
* Written informed consent

Exclusion Criteria:

* Known hypersensitivity/allergy to study products and/or materials used
* teeth having deep carious lesions or extensive restorations
* Unwillingness to be randomly assigned to 1 of the 3 treatment groups
* Advanced periodontal disease.

Ages: 14 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in White spot lesions dimension | 6 months: (Baseline, 1 week, 1 month, 3 months, 6 months)
  Quantified using computer-assisted analysis based on digital intraoral photographs

SECONDARY OUTCOMES:
change in lesion fluorescence | 6 months: (Baseline, 1 week, 1 month, 3 months, 6 months)
  evaluated using diode laser fluorescence device (Diagnodent)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria, Egypt